CLINICAL TRIAL: NCT06513312
Title: A Phase 2, Open-label, Multicenter, Randomized Study to Evaluate the Persistence, Safety, Acceptability, and Pharmacokinetics of Twice Yearly Long-acting Subcutaneous Lenacapavir for HIV Pre-Exposure Prophylaxis (PrEP) in People Who Would Benefit From PrEP
Brief Title: Study of Lenacapavir Taken Twice a Year for HIV Pre-Exposure Prophylaxis (PrEP)
Acronym: PURPOSE 5
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GS-US-528-6727; 2023-507891-31 (Other: EU CT Number)
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Pre-Exposure Prophylaxis of HIV Infection
MeSH Terms: interventions — lenacapavir; Emtricitabine; Tenofovir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Randomized Phase: Lenacapavir (LEN) Group (Experimental): Participants will receive subcutaneous (SC) LEN 927 mg on Day 1 and 26 weeks and oral LEN 600 mg on Day 1 and 2.
  Interventions: Drug: Lenacapavir Injection; Drug: Lenacapavir Tablet
- Randomized Phase: F/TDF (Active Comparator): Participants will receive daily F/TDF (200/300 mg) fixed dose combination (FDC) tablets for up to 52 weeks.
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate (F/TDF)
- LEN Open Label Extension (OLE) Phase (Experimental): Participants in the F/TDF group will transition to get LEN and participants in the LEN group will continue to get LEN. All participants will get SC LEN on Day 1 and week 26 of the OLE phase.
  Interventions: Drug: Lenacapavir Injection; Drug: Lenacapavir Tablet
- Pharmacokinetic (PK) Tail Phase: F/TDF (Experimental): After completion of the LEN OLE Phase or upon discontinuation from the Randomized Phase for those receiving LEN, participants will be transitioned to receive F/TDF in the PK Tail Phase. Participants will receive once daily F/TDF for 78 weeks, beginning 26 weeks after the last LEN injection
  Interventions: Drug: Emtricitabine/tenofovir disoproxil fumarate (F/TDF)

INTERVENTIONS:
Drug: Lenacapavir Injection — Administered subcutaneously
  Other Names: GS-6207; Yeztugo®
  Arms: LEN Open Label Extension (OLE) Phase; Randomized Phase: Lenacapavir (LEN) Group
Drug: Lenacapavir Tablet — Administered orally
  Other Names: GS-6207
  Arms: LEN Open Label Extension (OLE) Phase; Randomized Phase: Lenacapavir (LEN) Group
Drug: Emtricitabine/tenofovir disoproxil fumarate (F/TDF) — Administered orally
  Other Names: Truvada®
  Arms: Pharmacokinetic (PK) Tail Phase: F/TDF; Randomized Phase: F/TDF

SUMMARY:
The goals of this clinical study are to learn more about the study drug lenacapavir (LEN), by comparing the consistent and continuous use of LEN and emtricitabine/tenofovir disoproxil fumarate (coformulated; Truvada®) (F/TDF), then by observing the safety of LEN and F/TDF, evaluating the acceptability of LEN injections and oral F/TDF, and observe how LEN moves throughout the body in people who would benefit from pre-exposure prophylaxis (PrEP).

The primary objective of this study is to compare LEN and F/TDF consistent and continuous use among people who would benefit from PrEP.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to comprehend and provide a signed written informed consent, which must be obtained prior to initiation of study procedures.
* Cisgender men who have sex with men, transgender women, transgender men, cisgender women, and nonbinary people.
* Increased likelihood of HIV acquisition as indicated by at least one of the following:

  1. Condomless sex with ≥ 2 partners in the past 6 months
  2. Diagnosis of a bacterial sexually transmitted infection (STI) in the past 12 months
  3. Engagement in sex work or transactional sex in the past 12 months
  4. Use of ≥ 2 courses of nonoccupational HIV post-exposure prophylaxis (nPEP) in the past 12 months
  5. Condomless sex with a partner living with HIV who has unknown or unsuppressed viral load (≥ 200 copies/mL) in the past 12 months
* Negative local rapid HIV-1/2 antibody (Ab)/antigen (Ag) test, central HIV-1/2 Ab/Ag, and HIV-1 RNA quantitative nucleic acid amplification testing (NAAT) at screening.

  1) If rapid HIV-1/2 Ab/Ag tests are unavailable due to extenuating circumstances, sites may run a laboratory-instrumented HIV-1/2 Ab/Ag test at their local laboratory, only if they confirm this is a fourth-generation assay and the time from blood draw to injection at any injection visit is < 48 hours.
* Estimated glomerular filtration rate (GFR) at least 60 mL/min at screening according to the Cockcroft-Gault formula for creatinine clearance (CLcr):

  * (140 - age in years) × (weight in kg) x (0.85 if female) = CLcr (mL/min) / 72 × (serum creatinine in mg/dL)

Key Exclusion Criteria:

* Coenrollment in any other clinical study (including observational) without prior approval from the sponsor is prohibited while participating in this study.
* Known hypersensitivity to the study drug, the metabolites, or formulation excipient.
* Current use of PrEP, defined as the use of PrEP in the preceding 4 weeks. PrEP should not be discontinued to facilitate study participation. For cabotegravir, this is defined as 4 weeks since the next injection was due (ie, 12 weeks since their most recent cabotegravir injection).
* Current use of nPEP, unless the prescribed course will be completed prior to randomization.
* Past or current participation in HIV vaccine or HIV broadly neutralizing Ab study unless participant provides documentation of receipt of placebo (ie, not active product).
* Acute viral hepatitis A, B, or C or evidence of chronic hepatitis B or C infection
* Severe hepatic impairment or a history of or current clinical decompensated liver cirrhosis (eg, ascites, encephalopathy, variceal bleeding).
* Have a suspected or known active, serious infection(s) (eg, active tuberculosis, etc).

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender male, Cisgender female, Transgender male, Transgender female, and Gender non-binary
Enrollment: 268 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with LEN and F/TDF Persistence through 52 Weeks | Up to Week 52
  This outcome measure will compare LEN and F/TDF persistence through 52 weeks, where persistence is defined by On-time LEN Injection at Day 1/Baseline and Week 26 and On-time Follow-up Visit at Week 52 for LEN arm and by Adherence Levels Based on tenofovir diphosphate (TFV-DP) concentrations in red blood cells consistent with ≥ 4 doses/week (≥ 700 fmol/punch) in dried blood spot (DBS) at Weeks 13, 26, 39, and 52 for F/TDF arm.

SECONDARY OUTCOMES:
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose date up to 30 days post last dose at Week 78
Percentage of Participants Experiencing Treatment-emergent Clinical Laboratory Abnormalities | First dose date up to 30 days post last dose at Week 78
Overall acceptability of LEN and F/TDF as PrEP as Assessed by Percentage of Participants with responses to Question on Acceptability | Up to Week 52
  To assess the acceptability of the study drug, participants will complete the questionnaire including a question on general acceptability of the assigned study drug on an ordinal 5-category scale with a response of: Completely unacceptable, Unacceptable, No opinion, Acceptable, or Completely acceptable.
Pharmacokinetic (PK) Parameter: Ctrough for LEN at Week 26 | Week 26
  Ctrough is defined as the concentration at the end of the dosing interval.
PK Parameter: Ctrough for LEN at Week 52 | Week 52
  Ctrough is defined as the concentration at the end of the dosing interval.

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (14):
- France (6):
  - Hopital Avicenne, Bobigny
  - Hopital Europeen Marseille, Marseille
  - CHU Nice Archet, Nice
  - Hopital Saint Louis - Assistance Publique des Hopitaux de Paris, Paris
  - APHP Hopital Saint-Antoine, Paris
  - APHP Bichat Claude-Bernard Hospital, Paris
- United Kingdom (8):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham Heartlands Hospital, Birmingham
  - Clinical Research Facility, University Hospitals Sussex NHS Foundation Trust, Brighton
  - Axess Sexual Health, Liverpool University Hospitals NHS Trust, Liverpool
  - Grahame Hayton Unit, Ambrose King Centre, Royal London Hospital, Barts Health NHS Trust, London
  - Homerton Healthcare NHS Foundation Trust, Homerton University Hospital, London
  - Caldecot Centre, Kings College Hospital, Kings College Hospital NHS Foundation Trust, London
  - Chelsea and Westminster Hospital NHS Foundation Trust, Clinical Research Facility, Chelsea and Westminster Hospital, London
  - Manchester University NS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT06513312